CLINICAL TRIAL: NCT02445404
Title: Randomized Phase II Study to Compare Efficacy of CHOP Versus Fractionated ICED in Transplant-eligible Patients With Previously Untreated Peripheral T-cell Lymphoma
Brief Title: Compare Efficacy of CHOP Versus Fractionated ICED in Transplant-eligible Patients With Previously Untreated PTCL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Seog Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-12-011
Record Dates: First submitted 2015-05-12; First posted 2015-05-15 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Peripheral T-cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Cyclophosphamide; Vincristine; Prednisone; Ifosfamide; Carboplatin; Etoposide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CHOP (Active Comparator): cyclophosphamide, 750mg/m² IV day1 doxorubicin, 50 mg/m² IV day1 vincristine, 1.4 mg/m² (max 2 mg) IV day1 prednisone ,40 mg/m² PO day1~5 every 3 weeks
  Interventions: Drug: CHOP; Drug: fractionated ICED
- Fractionated ICED (Experimental): ifosfamide, 1.67 g/m² IV day1~3 carboplatin, AUC =5 IV day1 etoposide, 100mg/m² IV day1~3 dexamethasone 40 mg PO or IV day1~4 every 3 weeks
  Interventions: Drug: CHOP; Drug: fractionated ICED

INTERVENTIONS:
Drug: CHOP — cyclophosphamide, 750mg/m² IV day1 doxorubicin, 50 mg/m² IV day1 vincristine, 1.4 mg/m² (max 2 mg) IV day1 prednisone ,40 mg/m² PO day1~5 every 3 weeks
  Other Names: cyclophosphamide, cyclophosphamide, vincristine,prednisone
Drug: fractionated ICED — ifosfamide, 1.67 g/m² IV day1~3 carboplatin, AUC =5 IV day1 etoposide, 100mg/m² IV day1~3 dexamethasone 40 mg PO or IV day1~4 every 3 weeks
  Other Names: ifosfamide, carboplatin, etoposide, dexamethasone

SUMMARY:
This study is a Randomized Phase II Study to Compare Efficacy of CHOP versus Fractionated ICED in Transplant-eligible Patients with Previously Untreated Peripheral T-cell Lymphoma.

DETAILED DESCRIPTION:
It recommends that the CHOP regimen in the primary T-cell lymphoma therapies currently used but did not get satisfactory effect of therapy (progression-free survival 40%), primarily to consider the clinical trial at NCCN guideline.But why the CHOP regimen is widely used because physicians are accustomed to use. Fractionated ICED therapy is a therapy by adjusting the Original ICE regimen.This is how the capacity of Ifosfamide divided into three days. (Fractionated ifosfamide).Original ICE therapy has been widely used as a salvage therapy of patients with relapsed or refractory lymphoma for a long time, it has been recommended as part of primary therapy of T-cell lymphoma.But Fractionated ICED is added to dexamethasone therapy in order to improve the effectiveness as a primary therapy.The recurrent lymphoma in 75 patients with treatment after Fractionated ICE when the self-stem cell transplantation, showed a more than 40% progression-free survival.Thus treatment of Fractionated ICED targeting previously untreated patients, and if a combination of high-dose dexamethasone to expect to be able to induce a progression-free survival of 60% or more.

ELIGIBILITY:
Inclusion Criteria:

1. Age 19-65 years
2. Informed consent
3. Subject able to adhere to the study visit schedule and other protocol requirements.
4. Histologically proven Peripheral T-cell Lymphoma,No prior chemotherapy for the treatment of Peripheral T-cell Lymphoma It includes the following subtypes.

   * PTCL, not otherwise specified
   * Angioimmunoblastic T-cell lymphoma
   * Anaplastic large cell lymphoma, ALK-negative type
   * Enteropathy-associated T-cell lymphoma
   * Hepato-splenic T-cell lymphoma
   * Subcutaneous panniculitis-like T-cell lymphoma
   * Primary cutaneous gamma-delta T-cell lymphoma
   * Primary cutaneous CD8+ aggressive epidermotropic lymphoma
   * Other non classifiable T-cell Lymphoma
5. Performance status (ECOG) 0,1 or 2
6. A negative pregnancy test prior to treatment must be available both for pre-menopausal women
7. Female of childbearing potential (FCBP) must: contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) while on IP; and for 3 months following the last dose of IP.Male subjects must practice true abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions, and for 3 months following IP discontinuation.
8. life expectancy≥90day(3months)

Exclusion Criteria:

1. Other serious medical illnesses or psychiatric disorders
2. Any state that the confusion in the interpretation of test result.
3. Other type lymphoma ex) B-cell lymphoma
4. Other type T-cell lymphoma

   * Adult T-Cell Leukemia/Lymphoma
   * NK/T-cell Lymphoma, Nasal Type
   * ALK-Positive Anaplastic Large-Cell Lymphoma
   * Cutaneous Tcell lymphoma
   * primary cutaneous CD30+ lympho- proliferative disorder
   * primary cutaneous Anaplastic T cell lymphoma
5. Previously treated for PTCL(Except for a short period before randomization of corticosteroids (a period of not more than 8 days)
6. Previous radiation therapy
7. CNS involvement.
8. If the contraindication to chemoherapy
9. Subject has known historical or active infection with HIV.
10. BM function: ANC < 1.5 × 109/L; Platelet count <100,000/mm2 (100 × 109/L), SGOT/AST or SGPT/ALT ≥ 3.0 x ULN, Bilirubin> 2 x upper normal value
11. serum creatinine level > 2.0 x ULN
12. Any other malignancies within the past 3 years except curatively treated non-melanoma skin cancer or in situ carcinoma of cervix uteri
13. MUGA scan <45%
14. Those who administered doxorubicin exceeding 200 mg / m2
15. Subject has active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy.
16. Breast-feeding or pregnant female

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2015-09-23 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 3 years
  Time to disease progression is defined as the time from treatment start to the first recording of relapse or disease progression or death of any cause

SECONDARY OUTCOMES:
Overall survival | 3 years
  Duration of survival is defined as the time from treatment start to death of any cause or the date of last follow-up. Subjects who are alive will be censored using the date at which they are last known to be alive
overall response rate | 3 years
  They should be classified as complete remission(CR),Partial remission(PR),Stable disease(SD), or progression disease(PD)according to the Revised Response Criteria for Malignant Lymphoma
Response duration | 3 years
Toxicity profiles | 3 years
  Toxicity profiles as measured by Adverse Events and Laboratory results.

CONTACTS AND LOCATIONS:
Overall Officials: Won Seog Kim, MD,Ph.D., Principal Investigator — Samsung Medical Center,Seoul,Korea
Locations (1):
- Samsung Medical Center, Seoul, Seoul, Korea, Republic of, South Korea

IPD SHARING:
Plan to Share IPD: Undecided